CLINICAL TRIAL: NCT06964191
Title: A Phase 2 Randomized, Multi-center, Parallel, Active-controlled Clinical Study to Evaluate the Safety and Efficacy of Intracameral PA5108 Ocular Implants in Patients With Primary Open-angle Glaucoma, or Ocular Hypertension
Brief Title: Evaluate Efficacy and Safety of PA5108 Ocular Implants in Primary Open Angle Glaucoma or Ocular Hypertension
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PolyActiva Pty Ltd (Industry)
Collaborators: IUVO S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LATA-CS201
Record Dates: First submitted 2025-03-25; First posted 2025-05-09 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the study design, the product and the treatment arms, neither the study Investigator nor participant can be completely masked as to the treatment being administered. The participant will be aware of randomization to either an ocular implant or eye drops but will remain masked as to the strength of implant administered.
  The Investigator and implant administration personnel will be unmasked and be able to determine which strength of implant has been administered due to the size of the implant. Intraocular pressure assessments and certain safety assessments should be observer masked to the extent possible.
  Study personnel/technicians performing some study assessments will be masked to the treatment randomization to the extent possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PA5108 Ocular Implant low dose (Experimental): PA5108 Ocular Implant, low dose in the study eye, and latanoprost ophthalmic solution 0.005% once daily pm in the other eye.
  Interventions: Combination Product: PA5108 Ocular Implant low dose; Drug: Latanoprost 0.005% Ophthalmic Solution
- PA5108 Ocular Implant high dose (Experimental): PA5108 Ocular Implant, high dose in the study eye, and latanoprost ophthalmic solution 0.005% once daily pm in the other eye.
  Interventions: Combination Product: PA5108 Ocular Implant, high dose; Drug: Latanoprost 0.005% Ophthalmic Solution
- Latanoprost ophthalmic solution 0.005% (Active Comparator): Latanoprost ophthalmic solution 0.005% once daily pm in both eyes.
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution

INTERVENTIONS:
Combination Product: PA5108 Ocular Implant low dose — The PA5108 Ocular Implant low dose is supplied preloaded into the needle of a single use administration device ready for use.
  Arms: PA5108 Ocular Implant low dose
Combination Product: PA5108 Ocular Implant, high dose — The PA5108 Ocular Implant high dose is supplied preloaded into the needle of a single use administration device ready for use.
  Arms: PA5108 Ocular Implant high dose
Drug: Latanoprost 0.005% Ophthalmic Solution — Latanoprost eye drops at a concentration of 0.005%

SUMMARY:
The goal of this clinical trial is to determine the dose of PA5108 Ocular Implant that is effective and safe for the reduction of intraocular pressure in adult patients with open-angle glaucoma or ocular hypertension, compared to the standard treatment therapy.

DETAILED DESCRIPTION:
This is a randomised, parallel, masked, active-controlled study that will evaluate the efficacy and safety of a low dose and a high dose of PA5108 Ocular Implant with single redosing during the study, in adults with open-angle glaucoma or ocular hypertension.

The study will also collect information on the implant administration procedure and overall experience from study participants.

The study plans to recruit approximately 75 participants.

Eligible participants will be randomly selected to receive one of the following treatments:

* PA5108 Ocular Implant - low dose in the study eye, and Latanoprost 0.005% eye drops in the other eye
* PA5108 Ocular Implant - high dose in the study eye, and Latanoprost 0.005% eye drops in the other eye
* Latanoprost 0.005% eye drops in both eyes (control treatment group) If allocated to receive either of the ocular implants, a second implant of the same dose will be administered at 26 weeks and participants will be followed for safety and intraocular pressure control until week 58 or until the implant is no longer visible in the study eye.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to provide informed consent and follow study instructions
* 18 years of age or older
* Diagnosis of open-angle glaucoma or ocular hypertension in both eyes
* Qualifying IOPs across 2 visits following washout of IOP-lowering medication, if applicable
* Qualifying best-corrected visual acuity BCVA using Early Treatment Diabetic Retinopathy Study (ETDRS) chart in study eye
* Qualifying corneal endothelial cell density (CEDC) in the study eye

Key Exclusion Criteria:

* Pseudoexfoliation or pigment dispersion, narrow irido-corneal drainage angles, or existing peripheral anterior synechiae in the inferior angle either eye.
* Advanced or severe glaucoma
* Disqualifying central corneal thickness in either eye
* Significant other ocular conditions that could prevent accurate assessment of IOP and corneal health
* Uncontrolled medical conditions
* Have previously received, any injectable glaucoma medication into the anterior chamber of the study eye
* Have received intravitreal injections in the study eye within the last 3 months of the Screening Visit and anticipated need for an intravitreal injection during the course of the study
* Unwilling or unable to discontinue, in either eye, soft contact lens wear at least 2 days and hard contact lens wear 1 week before scheduled study visits and on implant administration days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy: change in mean diurnal intraocular pressure in study eye | From Baseline to 12 weeks
Incidence of ocular symptoms and ocular treatment-emergent adverse events. | Day 1 to study completion until at least Week 58
  Ocular safety and tolerability (AEs)
Clinically significant change on slit-lamp exam | Day 1 to study completion until at least Week 58
  Slit-lamp biomicroscopy of eye to observe clinically significant changes.
Clinically significant change in corneal endothelial cells | Day 1 to study completion until at least Week 58
  Corneal endothelial cell density (cells/mm2) measured by specular microscopy.

SECONDARY OUTCOMES:
Efficacy: intraocular pressure change from baseline in study eye at different diurnal time points. | Weeks 2-52

OTHER OUTCOMES:
Exploratory: Gather data on implant administration procedure and overall experience from study participants. | At 24 and 58 weeks
  A questionnaire comprising two questions will be used at Week 24 and Week 58 to assess the administration procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No